CLINICAL TRIAL: NCT02748486
Title: Efficacy of Metacognitive Training Single Modules: Jumping to Conclusions and To Empathize... Among Patients of Psychiatric Rehabilitation Ward With Diagnosis of Schizophrenia.
Brief Title: Efficacy of Metacognitive Training Single Modules: Jumping to Conclusions and To Empathize...
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warsaw (Other)
Collaborators: Medical University of Warsaw (Other); Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Principal Investigator, Joachim Kowalski, MSSc, University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BadaniaWłasne0001
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: schizophrenia; randomized controlled trial; metacognitive training; single sessions
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Jumping To Conculsions (Experimental): Metacognitive Training Jumping to conclusions module
  Interventions: Behavioral: Metacognitive Training Jumping to Conclusion
- Theory of Mind (Experimental): Metacognitive Training To empathize... module
  Interventions: Behavioral: Metacognitive Training To Empathize
- Control (Sham Comparator): group discussion of current events
  Interventions: Behavioral: Group discussion

INTERVENTIONS:
Behavioral: Metacognitive Training Jumping to Conclusion — Therapeutical intervention based on cognitive-behavioural therapy paradigm. Addresses cognitive bias of schizophrenia patients - jumping to conclusion.
  Arms: Jumping To Conculsions
Behavioral: Group discussion — Group discussion of current events
  Arms: Control
Behavioral: Metacognitive Training To Empathize — Therapeutical intervention based on cognitive-behavioural therapy paradigm. Addresses cognitive bias of schizophrenia patients - Theory of Mind deficits.
  Arms: Theory of Mind

SUMMARY:
The purpose of this study is to determine whether modules of Metacognitive Training: Jumping to Conclusions and To empathize... are effective in the treatment of patients with schizophrenia. Also it was investigated whether these modules have specific impact on cognitive biases severity.

DETAILED DESCRIPTION:
Investigators employ randomized controlled trial design. Patients in ward were recruited for the study in three waves. In each wave patients were assessed pre-intervention, then randomly allocated in one of three groups: with modules of Metacognitive Training or control group. Then patients were assessed post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of psychotic disorders
* informed consent

Exclusion Criteria:

* neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Fish Task | up to 3h after intervention
  variation of Beads Task used for measurement of jumping to conclusion
Reading the Mind in the Eyes Test | up to 3h after intervention
  used for measurement of Theory of Mind aspects
Cognitive Biases Questionnaire for Psychosis | up to 3h after intervention
  used for measurement of cognitive biases characteristic for psychotic patients

SECONDARY OUTCOMES:
Symptom Checklist 27 plus | up to 3h after intervention
  screening tool for psychopathology symptoms
Paranoia Checklist | up to 3h after intervention
  questionnaire used for assessment of paranoid ideation

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Gawęda, MD, Study Chair — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuncewicz D, Dragan M, Hardt J. [Validation of the Polish version of the symptom checklist-27-plus questionnaire]. Psychiatr Pol. 2014 Mar-Apr;48(2):345-58. Polish. PMID 25016771
- [Background] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Background] Moritz S, Woodward TS. Jumping to conclusions in delusional and non-delusional schizophrenic patients. Br J Clin Psychol. 2005 Jun;44(Pt 2):193-207. doi: 10.1348/014466505X35678. PMID 16004654
- [Background] Freeman D, Garety PA, Bebbington PE, Smith B, Rollinson R, Fowler D, Kuipers E, Ray K, Dunn G. Psychological investigation of the structure of paranoia in a non-clinical population. Br J Psychiatry. 2005 May;186:427-35. doi: 10.1192/bjp.186.5.427. PMID 15863749